CLINICAL TRIAL: NCT03267589
Title: NSGO-OV-UMB1; ENGOT-OV30 / NSGO: A Phase II Umbrella Trial in Patients With Relapsed Ovarian Cancer
Brief Title: Trial in Patients With Relapsed Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other)
Collaborators: Gynecologic Cancer Intergroup (GCIG) (Other); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENGOT-OV30 / NSGO
Record Dates: First submitted 2017-07-05; First posted 2017-08-30 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Ovarian Cancer
Keywords: immunotherapy; ovarian cancer; durvalumab; tremelilumab; MEDI 9447; MEDI 0562
MeSH Terms: conditions — Ovarian Neoplasms | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: Part 1: single cohorts of novel agents Part 2: randomized phase 2 against standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort A (Experimental): Intervention: MEDI9447 (CD73) + durvalumab
  Interventions: Drug: Durvalumab, Tremelilumab, MEDI 9447, MEDI 0562
- Cohort B (Experimental): Intervention: MEDI0562 (OX40) + durvalumab
  Interventions: Drug: Durvalumab, Tremelilumab, MEDI 9447, MEDI 0562
- Cohort C (Experimental): Intervention: MEDI0562 (OX40) + tremelimumab combination
  Interventions: Drug: Durvalumab, Tremelilumab, MEDI 9447, MEDI 0562

INTERVENTIONS:
Drug: Durvalumab, Tremelilumab, MEDI 9447, MEDI 0562 — Three different combination are being tested. Each cohort has different combination

SUMMARY:
The overall objectiv is to obtain preliminary evidence of efficacy of novel agents for the management of relapsed ovarian cancer, and in part 2 efficacy of novel agents compared to the standard of care (SoC).

ELIGIBILITY:
Inclusion Criteria:

1. Platinum-sensitive disease: defined as disease progression ≥ 6 months following the last administered dose of platinum-based therapy. Patients must have received atleast one line of chemotherapy for platinum-sensitive disease. OR
2. Platinum-resistant disease: defined as disease progression < 6 months following the last administered dose of platinum-based therapy.

   OR
3. Platinum-refractory disease: defined as lack of response or disease progression while receiving the most recent therapy.

   Other key inclusion criteria:
4. Histological confirmed ovarian, fallopian tube or peritoneal cancers.
5. Histological types: high-grade serious, high-grade endometriod, undifferentiated, carcinosarcoma or mixed histology.
6. Subjects must have at least 1 measurable lesion as defined by RECIST guidelines. This should not be the same lesion used for biopsy.
7. Patients entering cohort A: Archival tumour tissue must be screened for CD73 and only CD73 positive patients (defined as >10% of tumor cells positive) will enter this trial.
8. Patient agrees to undergo all analysis (blood, serum, tissue); radiological examinations according to protocol.
9. Mandatory tumour biopsy before treatment (before day 0) and at day 56 of treatment.
10. Patients must give informed consent.
11. Patients must be at least 18 years of age.
12. ECOG performance status 0-1
13. Serum albumin >30g/l.
14. Adequate organ function
15. Life expectancy of at least 12 weeks.
16. Patients must be fit to receive Investigational medical products (IMPs)

Exclusion Criteria:

1. Subjects using immunosuppressive medications within 14 days.
2. Immunodeficiency or organ transplant
3. Live vaccines within 28 days prior to the first dose.
4. Major surgery within 28 days prior to the first dose.
5. Ovarian sarcomas, small cell carcinoma with neuroendocrine differentiation, non-epithelial can-cers.
6. Cancer therapies (chemotherapy, radiotherapy, surgery, immunotherapy, biologic or hormonal therapy) within 28 days prior to the first dose.
7. Concurrent treatment with an investigational agent or participation in another clinical trial.
8. Previous malignant disease: patients are not eligible for the study if actively being treated of inva-sive cancer other than ovarian cancer. Patients with previous malignant disease other than ovarian cancer who are relapse-free and treatment-free for more than three years may enter this study. Pa-tients with previous history of in-situ carcinoma, stage 1A cervical cancer or non-invasive basal cell and squamous cell skin carcinoma can enter this trial.
9. Active infection including tuberculosis
10. History of a cerebral vascular accident, transient ischemic attack or subarachnoid hemorrhage within the past 6 months.
11. History of clinically significant hemorrhage in the past 3 months.
12. Untreated CNS disease, leptomeningeal disease or cord compression. Subjects with treated dis-ease should have at least 4 weeks of neurologic and radiographic stability and be off steroids for 14 days.
13. Significant cardiovascular disease's.
14. Persistance of clinically relevant therapy related toxicity from previous anticancer therapy (any grade 3-4 toxicity or grade ≥2 neuropathy).
15. Known hypersensitivity to the trial drugs, or to their excipients.
16. Has had prior exposure to IMPs, or any other immunotherapy.
17. Active or prior documented autoimmune or inflammatory disorders
18. For cohorts B and C: Medical condition requiring current systemic anticoagulation, or a history of congenital hypercoagulable condition. Subjects taking aspirin at doses < 325 mg per day are eli-gible provided that prothrombin time is within the institutional range of normal. Use of local anti-coagulation for port maintenance is permitted

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
Disease control rate (DCR) | 16 weeks
  Disease control rate (DCR) (CR+PR+SD)

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) by RECIST v1.1 | 10 months
  PFS by RECIST v1.1
PFS by Immune-RECIST | 10 months
  PFS by Immune-RECIST
Overall survival (OS) | 36 months
  Overall survival (OS)
Objective response rate | 10 months
  Objective response rate according to RECIST v1.1 (ORR)
Duration of (Overall) Response (DoR) | 10 months
  Duration of (Overall) Response (DoR)

CONTACTS AND LOCATIONS:
Overall Officials: Mansoor R Mirza, MD, Study Director — NSGO-CTU
Locations (5):
- Denmark (2):
  - Rigshospitalet, København Ø, Region Sjælland
  - VejleSygehus, Vejle, Region Syddanmark
- Tampere University Hospital, Tampere, Finland
- Norway (2):
  - Haukeland University Hospital, Bergen, Haukeland
  - The Norwegian Radium Hospital, Oslo

IPD SHARING:
Plan to Share IPD: Yes
Upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From December 2023.